CLINICAL TRIAL: NCT00834873
Title: A Randomized, Two-Way Crossover, Single-Dose, Open Label Study to Evaluate the Relative Bioavailability of a Test Tablet Formulation of Carvedilol (25 mg), Compared to an Equivalent Dose of COREG® (SmithKline Beecham Pharmaceuticals) in 24 Fed, Healthy, Adult Subjects
Brief Title: Carvedilol (25 mg) in 24 Fed, Healthy, Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 01269
Record Dates: First submitted 2009-01-30; First posted 2009-02-03 (Estimated); Results first posted 2009-08-18 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Experimental): Carvedilol 25 mg Tablet (test) dosed in first period followed by Coreg® 25 mg Tablet (reference) dosed in second period
  Interventions: Drug: Carvedilol 25 mg tablets
- Coreg® (Active Comparator): Coreg® 25 mg Tablet (reference) dosed in first period followed by Carvedilol 25 mg Tablet (test) dosed in second period
  Interventions: Drug: COREG® 25 mg tablets

INTERVENTIONS:
Drug: Carvedilol 25 mg tablets — 1 x 25 mg
  Arms: Carvedilol
Drug: COREG® 25 mg tablets — 1 x 25 mg
  Arms: Coreg®

SUMMARY:
The objective of this randomized, single-dose, two-way crossover evaluation is to compare the relative bioequivalence of a test carvedilol formulation (TEVA Pharmaceuticals USA) to and equivalent oral dose of the commercially available carvedilol (COREG®, SmithKline Beecham Pharmaceuticals) in a test population of 24 adult individuals under fed conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Sex: Male of Female; similar proportions of each preferred.
* Age: At least 18 years.
* Weight: Minimum of 120 pounds and a BMI (body mass index) of less than 30.

Exclusion Criteria:

* Subjects not complying with the above inclusion criteria must be excluded from the study.
* In addition, any one of the conditions listed below will exclude a subject from the study.
* History of treatment for alcoholism, substance abuse, or drug abuse within the past 24 months
* History of malignancy, stroke, diabetes, cardiac, renal or liver disease, or other serious illness.
* History of treatment for any gastrointestinal disorder within the past five (5) years.
* History of, or presence of, asthma
* History of peripheral vascular disease
* History of heart failure
* History of pre-existing cardiac arrythmias associated with tachycardia
* History of severe sensitivity to allergens, requiring urgent medical treatment.
* Females who are pregnant or lactating
* History of hypersensitivity to carvedilol, or any beta adrenergic blocking drug.
* Conditions upon screening which might contraindicate or require that caution be used in the administration of carvedilol, including:
* sitting systolic blood pressure below 100 mmHg, or diastolic pressure below 60 mmHg.
* Heart rate less than 60 beats per minute after a 5-minute rest in a seated position.
* Inability to read and/or sign the consent form.
* Treatment with any other investigational drug during the four (4) weeks prior to the initial dosing for this study.
* Subjects who smoke or use tobacco products or are currently using nicotine products (patches, gums,etc.) Ninety (90) days abstinence is required.
* subjects who have donated blood within four (4) weeks prior to the initial dosing for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-12; Primary Completion 2001-12 (Actual); Study Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M David Ayra, M.D., Principal Investigator — Gateway
Locations (1):
- Gateway Medical Research, Inc., Saint Charles, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Carvedilol (Test) First: Carvedilol 25 mg Tablet (test) dosed in first period follwed by Coreg® 25 mg Tablet (reference) dosed in second period
- Coreg® (Reference) First: Coreg® 25 mg Tablet (reference) dosed in first period followed by Carvedilol 25 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Carvedilol (Test) First | Coreg® (Reference) First
Started | 12 | 12
Completed | 12 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Washout: 7 Days
Arm/Group | Carvedilol (Test) First | Coreg® (Reference) First
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Carvedilol (Test) First | Coreg® (Reference) First
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Carvedilol (Test) First | Coreg® (Reference) First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 7 | 7 | 14
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasion | 11 | 9 | 20
  Black | 1 | 3 | 4
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration - Carvedilol in Plasma
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 60 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Carvedilol: Carvedilol 25 mg Tablet (test) dosed in either period
- Coreg®: Coreg® 25 mg Tablet (reference) dosed in either period
Arm/Group | Carvedilol | Coreg®
Number analyzed (Participants) | 23 | 23
ng/mL | 89.91 (40.86) | 97.05 (49.61)
Statistical Analysis 1: Comparison: Carvedilol vs Coreg®; Test type: Non-Inferiority or Equivalence — Using GLM procedures in SAS, analysis of variance (ANOVA)was performed on log-transformed AUC0-t, AUC0-inf and Cmax at the significance level of 0.05; Test/Ref Ratio of LS Means x 100 = 94.77, 90% CI [85.04 to 105.61] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated) - Carvedilol in Plasma
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 60 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Carvedilol | Coreg®
Number analyzed (Participants) | 23 | 23
ng*h/mL | 467.57 (287.12) | 490.16 (337.58)
Statistical Analysis 1: Comparison: Carvedilol vs Coreg®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 96.23, 90% CI [90.59 to 102.23] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant) - Carvedilol in Plasma
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 60 hour period
Population: Data from all subjects who completed the study were included in the statistical analysis.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Carvedilol | Coreg®
Number analyzed (Participants) | 23 | 23
ng*h/mL | 455.91 (284.99) | 478.61 (336.07)
Statistical Analysis 1: Comparison: Carvedilol vs Coreg®; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Test/Ref Ratio of LS Means x 100 = 96.11, 90% CI [90.45 to 102.12] — Bioequivalence is established when 90% Confidence Interval falls within 80 - 125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.